CLINICAL TRIAL: NCT04414020
Title: Cytoprotective Effect and Clinical Outcome of Perioperative Proesterone in Brain Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Principle investigator, Ministry of Health and Population, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 623-4/2020
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Diffuse Traumatic Cerebral Edema
Keywords: Progesterone; brain tumor; Neuronal biopsy
MeSH Terms: conditions — Brain Neoplasms | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Control group receiving conventional treatment without progesterone
- progesterone group (Active Comparator): 1mg pregesterone intramusculer given 7 days pre and post operative , Biopsy was achieved from brain tumor interface
  Interventions: Drug: Progesteron

INTERVENTIONS:
Drug: Progesteron — intramusculer progesterone
  Arms: progesterone group

SUMMARY:
Neuronal injury is evident in elective craniotomy for space occupying lesions. Surgical trauma and mechanichal impact of the tumor causes neuronal injury. Neurosreroid progesterone is a neurotransmittern , trail to use in abolishing neurotoxcicty

DETAILED DESCRIPTION:
Progesterone is a natural neurosteroid that we are trying to use to impede both direct neuronal injury cauesd by and indirectly by surgical trauma. Progesterone can decreas vasogenic brain oedema. Our primary outcome is to ameliorate microscopic cytoplasmic injury and decrease brain oedema exploited by biopsy from brain tumor interface. Exclusion criteria demonstratd as refusal to participate in the trial , emergency craniotomy, recurrent brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* All elective brain tumors elligible for craniotomy

Exclusion Criteria:

* Refusal to participare
* Emergency craniotomy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With craniotomy-Related Adverse Events | 3 months
  Degree of microscopic cellular injury and brain odema in brain biopsy

SECONDARY OUTCOMES:
Number of Participants with neuronal deficit | 2 months
  Sensory, motor or autonomic dysfunction

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Al Minyā, Abohelal
  - Faculty of Medicine, Minya, Abohelal

IPD SHARING:
Plan to Share IPD: No